CLINICAL TRIAL: NCT06365658
Title: Cognitive Functioning Profiles in Adults With Neurologically Recognized Aphasic Syndromes and General Population From a Biopsychosocial Perspective
Brief Title: Cognitive Functioning in Adults With Somatic Diseases and General Population From a Biopsychosocial Perspective
Status: Recruiting | Type: Observational
Sponsor: Bartosz M. Radtke (Other Government)
Responsible Party: Sponsor-Investigator, Bartosz M. Radtke, CEO, Laboratory of Psychological and Educational Tests
Organization: Laboratory of Psychological and Educational Tests (Other Government)
Other Study IDs: 2024/PTPiP/1
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Aphasia; Development, Human; Neuropathology
Keywords: aphasia; memory; learning; language; adults; seniors
MeSH Terms: conditions — Aphasia; Language

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- General population/control group: Polish adults (age 18 to 60 y.o).
  Interventions: Diagnostic Test: Psychological assessment
- Neurologically recognized aphasic syndromes: Polish adults (age 18 to 60 y.o) with neurologically recognized aphasic syndromes.
  Interventions: Diagnostic Test: Psychological assessment
- Seniors (over 60 y.o): Polish adults (over 60 y.o.)
  Interventions: Diagnostic Test: Psychological assessment

INTERVENTIONS:
Diagnostic Test: Psychological assessment — Psychological assessment of memory, learning and language

SUMMARY:
The goal of this observational study is to investigate cognitive functioning profiles in adults with neurologically recognized aphasic syndromes and general population.

The study group consist of minimal 600 adults (over 18 y.o.) who will be examined by qualified diagnosticians. Participants will be evaluated with tasks related to the studied variables: memory, learning and language. Furthermore informations regarding past and present health condition will be collected from participants.

The main questions it aims to answer are:

1. What is the profile of memory and learning among polish adults?
2. Do gender and age moderates patterns of memory and learning functioning among polish adults?
3. What is a specific pattern of language functioning in adults with neurologically recognized aphasic syndromes?
4. Do gender moderates specific patterns of language functioning in adults with neurologically recognized aphasic syndromes?

Researchers will compare the following groups of adults:

1. general population/control group
2. with neurologically recognized aphasic syndromes
3. seniors (over 60 y.o.)

ELIGIBILITY:
Inclusion criteria for general population/control group:

* age from 18 to 60 y.o.

Inclusion criteria for neurologically recognized aphasic syndromes

* age above 18 y.o.
* neurologically recognized aphasic syndromes

Inclusion criteria for seniors:

* age above 60 y.o.

Exclusion criteria for general population/control group:

* age less then 18 y.o.
* neurologically recognized aphasic syndromes

Exclusion criteria for neurologically recognized aphasic syndromes

* age less then 18 y.o.
* no neurologically recognized aphasic syndromes

Exclusion criteria for seniors

* age less then 60 y.o.
* diseases of the nervous system, such as: stroke, craniocerebral trauma, neuroinfections, neurodegenerative diseases
* mental disorders such as depression, psychotic disorders, anxiety disorders, addictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Polish adults.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-07-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Memory and learning | July 3, 2023 until June 30, 2026
  Test of Memory and Learning (second edition). A standardized test measuring memory functioning and learning abilities. The test includes four basic factors (Verbal Memory, Nonverbal Memory, Complex Memory, and Delayed Recall) and five supplementary factors (Attention/Concentration, Sequential Memory, Free Recall, Associative Recall and Learning). The raw scores obtained in each tested subscale are converted into scores scaled based on age norms, ranging from 1 to 20, where a higher score means better functioning of the examined area, and a lower result means poorer functioning.
Language | July 3, 2023 until June 30, 2026
  Boston Diagnostic Aphasia Examination-Third Edition. A spectrum of tools that helps to identify and distinguish among disorders of language function and neurologically recognized aphasic syndromes. The test have five functional subsections: 1) Conversational and Expository Speech, 2) Auditory Comprehension, 3) Oral Expression, 4) Reading and 5) Writing. The raw scores obtained in each tested subscale are converted into a percentile scale, ranging from 1 to 100, where a higher score means better functioning of the examined area, and a lower result means poorer functioning.
Socio-demographic data | July 3, 2023 until June 30, 2026
  Author's survey of socio-demographic data, including: gender, month and year of birth, region of residence

SECONDARY OUTCOMES:
General mental state | July 3, 2023 until June 30, 2026
  Mini-Mental State Examination. A clinical scale used to examine disorders in a patient's cognitive functioning. The questionnaire consists a series of questions allowing the assessment of the following functions: 1) orientation in time and place, 2) attention/concentration, 3) short-term memory (recall), 4) language skills, 5) visual-spatial abilities, 6) ability to understand and follow the instructions. The maximum score that can be obtained on the test is 30 points. 27-30 is a correct result; 24-26 is a cognitive impairment without dementia; 19-23 mean mild dementia; 11-18 is a moderate degree dementia and 0-10 mean profound dementia.
Health related data | July 3, 2023 until June 30, 2026
  Author's survey of health related data, including: hearing, eyesight, hypertension, atherosclerosis, previous heart attack, diabetes, endocrine diseases, respiratory system diseases, musculoskeletal system diseases, nervous system diseases, kidney diseases, sleep disorders, hospitalizations, procedures under general anesthesia, cancer, medications.
Education data | July 3, 2023 until June 30, 2026
  Author's survey of education, including: years of education, level of education, occupation, level of education of the participant's parents.

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Sajewicz-Radtke, Ph.D., Study Director — Laboratory of Psychological and Educational Tests; Bartosz M Radtke, Ph.D., Principal Investigator — Laboratory of Psychological and Educational Tests; Ariadna Łada-Maśko, Ph.D., Principal Investigator — Laboratory of Psychological and Educational Tests
Locations (1):
- Laboratory of Psychological and Educational Tests, Gdansk, Pomeranian Voivodeship, Poland